CLINICAL TRIAL: NCT03241355
Title: Double-blind, Parallel, Randomized, (Placebo-controlled) Explorative Study on the Effect of a Mixture of Prebiotic Oligosaccharides on the Composition of Intestinal Microbiota and Selected Health Outcomes in Children 3 to 6 Years of Age
Brief Title: Prebiotic Fructans on the Incidence of Acute Infectious Diseases in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beneo-Institute (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 13004n_Fructan_Study
Record Dates: First submitted 2017-08-03; First posted 2017-08-07 (Actual); Last update posted 2018-08-28 (Actual); Status verified 2018-08

CONDITIONS: Infectious Disease; Children, Only; Diet Modification
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- prebiotic inulin-type fructan (Active Comparator)
  Interventions: Dietary Supplement: prebiotic inulin-type fructan
- placebo maltodextrin (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo maltodextrin

INTERVENTIONS:
Dietary Supplement: prebiotic inulin-type fructan
  Arms: prebiotic inulin-type fructan
Dietary Supplement: Placebo maltodextrin
  Arms: placebo maltodextrin

SUMMARY:
The study aims to explore whether prophylactic dietary supplementation with prebiotic inulin-type fructans is able to influence the intestinal microbiota and the frequency of infectious disease episodes in kindergarten children during a winter period.

ELIGIBILITY:
Inclusion Criteria:

* Subject is healthy at the time of pre-examination
* Subject is aged 3-6 years at the time of pre-examination
* Subject attends a kindergarten at the time of pre-examination

Exclusion Criteria:

* congenital disease or malformation influencing the gastrointestinal System
* children with congenital or acquired immunodeficiency
* children with food intolerance, food allergy or metabolic disorder requiring special diet
* children who regularly (more than 3 times per week) consumed products or food supplements containing prebiotics or probiotics
* children who consumed antibiotics or laxatives within 14 days
* children who had any infectious disease within 14 days at the time of pre-examination

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 258 (Actual)
Dates: Start 2013-09-16 (Actual); Primary Completion 2014-04-28 (Actual); Study Completion 2014-04-28 (Actual)

PRIMARY OUTCOMES:
Frequency of infectious disease episodes | 24 weeks period

SECONDARY OUTCOMES:
microbiota composition | 24 weeks period
  fecal microbiota composition (qPCR, illumina)

CONTACTS AND LOCATIONS:
Overall Officials: Tamás Decsi, Prof., Principal Investigator — Department of Paediatrics, University of Pécs, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lohner S, Kullenberg D, Antes G, Decsi T, Meerpohl JJ. Prebiotics in healthy infants and children for prevention of acute infectious diseases: a systematic review and meta-analysis. Nutr Rev. 2014 Aug;72(8):523-31. doi: 10.1111/nure.12117. Epub 2014 Jun 5. PMID 24903007
- [Result] Lohner S, Jakobik V, Mihalyi K, Soldi S, Vasileiadis S, Theis S, Sailer M, Sieland C, Berenyi K, Boehm G, Decsi T. Inulin-Type Fructan Supplementation of 3- to 6-Year-Old Children Is Associated with Higher Fecal Bifidobacterium Concentrations and Fewer Febrile Episodes Requiring Medical Attention. J Nutr. 2018 Aug 1;148(8):1300-1308. doi: 10.1093/jn/nxy120. PMID 29982534
- [Derived] Soldi S, Vasileiadis S, Lohner S, Uggeri F, Puglisi E, Molinari P, Donner E, Sieland C, Decsi T, Sailer M, Theis S. Prebiotic supplementation over a cold season and during antibiotic treatment specifically modulates the gut microbiota composition of 3-6 year-old children. Benef Microbes. 2019 Apr 19;10(3):253-263. doi: 10.3920/BM2018.0116. Epub 2019 Feb 19. PMID 30776899